CLINICAL TRIAL: NCT06424119
Title: Multi-Center Randomized Study of Clinical and Inflammatory Outcomes in Intensive Cardiac Rehabilitation and Traditional Cardiac Rehabilitation Programs (CREDIBLE Study)
Brief Title: Multi-Center Study of Clinical and Inflammatory Outcomes in Intensive Cardiac Rehabilitation and Traditional Cardiac Rehabilitation Programs
Acronym: CREDIBLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pritikin ICR (Other)
Collaborators: Ballad Health (Other); Mission Health System, Asheville, NC (Other); Trinity Health System (Industry); Connecting Health Innovation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CREDIBLE
Record Dates: First submitted 2024-05-12; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Cardiovascular Diseases
Keywords: Intensive Cardiac Rehabilitation; Traditional Cardiac Rehabilitation
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: ICR-eligible patients are randomized into one of three groups of 150 patients: (1) ICR 72 session program with C2life® supplied food, (2) ICR 72 session without C2life® supplied food, or (3) TCR 36 session program without C2life supplied food (ICR-food, ICR-no food, and TCR-no food).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ICR-No Food (Experimental): Intensive Cardiac Rehab (ICR) 72-session program without C2life® supplied food
  Interventions: Behavioral: Intensive Cardiac Rehabilitation
- ICR-Food (Experimental): Intensive Cardiac Rehab (ICR_ 72-session program with C2life® supplied food
  Interventions: Behavioral: Intensive Cardiac Rehabilitation; Other: C2life® Food
- TCR-No Food (Active Comparator): Traditional Cardiac Rehab (TCR) 36-session program without C2life® supplied food
  Interventions: Behavioral: Traditional Cardiac Rehabilitation

INTERVENTIONS:
Behavioral: Traditional Cardiac Rehabilitation — Patient must have a qualifying cardiovascular event and eligible for ICR. Once patient is randomized to TCR arm, they will attend 36 sessions of the program at one of three locations.
  Other Names: TCR
  Arms: TCR-No Food
Behavioral: Intensive Cardiac Rehabilitation — Patient must have a qualifying cardiovascular event and eligible for ICR. Once patient is randomized to ICR arm, they will attend 72 sessions of the program at one of three locations.
  Other Names: ICR
  Arms: ICR-Food; ICR-No Food
Other: C2life® Food — Patient must have a qualifying cardiovascular event and eligible for ICR. Once patient is randomized to ICR arm with food, they will receive the food at the beginning of the second week of their respective program. Food will be delivered by mail weekly for a total of 11 weeks to the patient's home address.
  Arms: ICR-Food

SUMMARY:
The goal of this prospective study is to evaluate whether the Intensive Cardiac Rehabilitation (ICR) program provides incremental benefits over the Traditional Cardiac Rehabilitation (TCR) program, defined by readmission costs. The study aims to confirm:

* That ICR is associated with better outcomes than TCR, defined as lower readmission costs, lower incidence of major adverse cardiovascular events (MACE), and improvement in biomarkers, epigenetic markers, and inflammatory markers.
* The addition of food to the ICR program will further improve these outcomes.

ICR-eligible participants

* Will be randomized into one of three groups: (1) ICR 72 session program with home-delivered C2life® supplied food, (2) ICR 72 session without C2life® supplied food, or (3) TCR 36 session program without C2life supplied food
* Biometric measurements and laboratory measurements will be performed at entry into the rehab intervention, discharge from rehab intervention, and at 6 months after discharge.
* Epigenetic measurements will be performed at admission and discharge from the rehab intervention

ELIGIBILITY:
Inclusion Criteria:

* All patients eligible for an Intensive Cardiac Rehabilitation (ICR) Program at each of the three study sites outline below, stratified by one of the following qualifying cardiovascular events, including myocardial infarction (STEMI and NSTEMI), angioplasty and stents, coronary artery bypass, surgical or percutaneous valve repair or replacement, and stable congestive heart failure with reduced ejection fraction of 35% or less.

Exclusion Criteria:

* Anticipated life expectancy of under 2 years
* Any co-morbidity that would limit participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Readmission Rate Data | Followup may extend up to 5 years for a post-hoc EMR analysis.
  Readmission rate data will include:
  1. Actual number of all cause readmissions
  2. Days in hospital for each readmission
  3. Cost of readmission.
  Stratification between all cause and cardiovascular readmissions will be performed as an additional sub-analysis.

SECONDARY OUTCOMES:
MACE | At 1 and 2 years.
  MACE is defined as all-cause death, non-fatal MI, hospitalization for unstable angina, PCI, CABG, peripheral artery revascularization, Ischemic stroke, CHF hospitalization, heart valve surgery, and heart transplant.
Composite Total Readmission Rates | At 1 and 2 years
  Number of readmissions within 2 years.
Readmission Days | At 1 and 2 years
  Composite length of stay in days for the total readmission events and each MACE category within 2 years.
Dietary Inflammation Index (DII) | At admission, discharge from program (about 12 weeks), and 6 month post-discharge
  Scores will be calculated for the C2life® diet as a whole and for each participant at the prespecified measurement times.
Labs | At admission, discharge (about 12 weeks), and 6 months post-discharge
  Labs will include lipids, comprehensive metabolic profile, HbA1c, Hs-CRP, IL-6, TNF-alpha, IFN-gamma, and ceramides.
Epigenetic Biomarkers Performed by Prosper eDNA® | Buccal swab at admission and discharge (about 12 weeks)
  Buccal swab samples will be taken to obtain this data. We propose to use a set of epigenetic biomarkers to measure biological age, metabolic health, inflammation, and overall fitness.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Asbill, MD, Principal Investigator — Mission Health; David Beckner, MD, Principal Investigator — Ballad Health; Frank A. Smith, MD, Principal Investigator — Trinity Health System; James R. Hebert, ScD, MSPH, Principal Investigator — Connecting Health Innovations, LLC (CHI)
Locations (3):
- United States (3):
  - Trinity Health Ann Arbor, Ypsilanti, Michigan
  - Mission Health, Asheville, North Carolina
  - Ballad CVA Heart Institute, Kingsport, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Writing Group Members; Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, Das SR, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Isasi CR, Jimenez MC, Judd SE, Kissela BM, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Magid DJ, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Rosamond W, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee; Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2016 Update: A Report From the American Heart Association. Circulation. 2016 Jan 26;133(4):e38-360. doi: 10.1161/CIR.0000000000000350. Epub 2015 Dec 16. No abstract available. PMID 26673558
- [Background] Leon AS, Franklin BA, Costa F, Balady GJ, Berra KA, Stewart KJ, Thompson PD, Williams MA, Lauer MS; American Heart Association; Council on Clinical Cardiology (Subcommittee on Exercise, Cardiac Rehabilitation, and Prevention); Council on Nutrition, Physical Activity, and Metabolism (Subcommittee on Physical Activity); American association of Cardiovascular and Pulmonary Rehabilitation. Cardiac rehabilitation and secondary prevention of coronary heart disease: an American Heart Association scientific statement from the Council on Clinical Cardiology (Subcommittee on Exercise, Cardiac Rehabilitation, and Prevention) and the Council on Nutrition, Physical Activity, and Metabolism (Subcommittee on Physical Activity), in collaboration with the American association of Cardiovascular and Pulmonary Rehabilitation. Circulation. 2005 Jan 25;111(3):369-76. doi: 10.1161/01.CIR.0000151788.08740.5C. PMID 15668354
- [Background] McMahon SR, Ades PA, Thompson PD. The role of cardiac rehabilitation in patients with heart disease. Trends Cardiovasc Med. 2017 Aug;27(6):420-425. doi: 10.1016/j.tcm.2017.02.005. Epub 2017 Feb 15. PMID 28318815
- [Background] Kotseva K, Wood D, De Bacquer D; EUROASPIRE investigators. Determinants of participation and risk factor control according to attendance in cardiac rehabilitation programmes in coronary patients in Europe: EUROASPIRE IV survey. Eur J Prev Cardiol. 2018 Aug;25(12):1242-1251. doi: 10.1177/2047487318781359. Epub 2018 Jun 6. PMID 29873511
- [Background] Anderson L, Oldridge N, Thompson DR, Zwisler AD, Rees K, Martin N, Taylor RS. Exercise-Based Cardiac Rehabilitation for Coronary Heart Disease: Cochrane Systematic Review and Meta-Analysis. J Am Coll Cardiol. 2016 Jan 5;67(1):1-12. doi: 10.1016/j.jacc.2015.10.044. PMID 26764059
- [Background] Balady GJ, Williams MA, Ades PA, Bittner V, Comoss P, Foody JM, Franklin B, Sanderson B, Southard D; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee, the Council on Clinical Cardiology; American Heart Association Council on Cardiovascular Nursing; American Heart Association Council on Epidemiology and Prevention; American Heart Association Council on Nutrition, Physical Activity, and Metabolism; American Association of Cardiovascular and Pulmonary Rehabilitation. Core components of cardiac rehabilitation/secondary prevention programs: 2007 update: a scientific statement from the American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee, the Council on Clinical Cardiology; the Councils on Cardiovascular Nursing, Epidemiology and Prevention, and Nutrition, Physical Activity, and Metabolism; and the American Association of Cardiovascular and Pulmonary Rehabilitation. Circulation. 2007 May 22;115(20):2675-82. doi: 10.1161/CIRCULATIONAHA.106.180945. Epub 2007 May 18. PMID 17513578
- [Background] R. James Barnard, Ph.D. The Pritikin Program: Understanding its value in Preventing and Controlling common diseases
- [Background] Gomez-Delgado F, Katsiki N, Lopez-Miranda J, Perez-Martinez P. Dietary habits, lipoprotein metabolism and cardiovascular disease: From individual foods to dietary patterns. Crit Rev Food Sci Nutr. 2021;61(10):1651-1669. doi: 10.1080/10408398.2020.1764487. Epub 2020 Jun 9. PMID 32515660
- [Background] Wong MMH, Louie JCY. A priori dietary patterns and cardiovascular disease incidence in adult population-based studies: a review of recent evidence. Crit Rev Food Sci Nutr. 2022;62(22):6153-6168. doi: 10.1080/10408398.2021.1897517. Epub 2021 Mar 10. PMID 33715546
- [Background] Zhong VW, Ning H, Van Horn L, Carnethon MR, Wilkins JT, Lloyd-Jones DM, Allen NB. Diet Quality and Long-Term Absolute Risks for Incident Cardiovascular Disease and Mortality. Am J Med. 2021 Apr;134(4):490-498.e24. doi: 10.1016/j.amjmed.2020.08.012. Epub 2020 Sep 14. PMID 32941845
- [Background] Kiecolt-Glaser JK. Stress, food, and inflammation: psychoneuroimmunology and nutrition at the cutting edge. Psychosom Med. 2010 May;72(4):365-9. doi: 10.1097/PSY.0b013e3181dbf489. Epub 2010 Apr 21. PMID 20410248
- [Background] Shivappa N, Godos J, Hebert JR, Wirth MD, Piuri G, Speciani AF, Grosso G. Dietary Inflammatory Index and Cardiovascular Risk and Mortality-A Meta-Analysis. Nutrients. 2018 Feb 12;10(2):200. doi: 10.3390/nu10020200. PMID 29439509
- [Background] Mazidi M, Shivappa N, Wirth MD, Hebert JR, Mikhailidis DP, Kengne AP, Banach M. Dietary inflammatory index and cardiometabolic risk in US adults. Atherosclerosis. 2018 Sep;276:23-27. doi: 10.1016/j.atherosclerosis.2018.02.020. Epub 2018 Feb 15. PMID 30015256
- [Background] Marx W, Veronese N, Kelly JT, Smith L, Hockey M, Collins S, Trakman GL, Hoare E, Teasdale SB, Wade A, Lane M, Aslam H, Davis JA, O'Neil A, Shivappa N, Hebert JR, Blekkenhorst LC, Berk M, Segasby T, Jacka F. The Dietary Inflammatory Index and Human Health: An Umbrella Review of Meta-Analyses of Observational Studies. Adv Nutr. 2021 Oct 1;12(5):1681-1690. doi: 10.1093/advances/nmab037. PMID 33873204
- [Background] Asadi Z, Yaghooti-Khorasani M, Ghazizadeh H, Sadabadi F, Mosa-Farkhany E, Darroudi S, Shabani N, Kamel-Khodabandeh A, Bahrami A, Khorrami-Mohebbseraj MS, Heidari-Bakavoli S, Heidari-Bakavoli A, Esmaily H, Moohebati M, Oladi MR, Shivappa N, Hebert JR, Ferns GA, Ghayour-Mobarhan M. Association between dietary inflammatory index and risk of cardiovascular disease in the Mashhad stroke and heart atherosclerotic disorder study population. IUBMB Life. 2020 Apr;72(4):706-715. doi: 10.1002/iub.2172. Epub 2019 Oct 16. PMID 31617677
- [Background] Todendi PF, Salla R, Shivappa N, Hebert JR, Ritter J, Cureau FV, Schaan BD. Association between dietary inflammatory index and cardiometabolic risk factors among Brazilian adolescents: results from a national cross-sectional study. Br J Nutr. 2022 Aug 28;128(4):744-752. doi: 10.1017/S0007114521003767. Epub 2021 Sep 21. PMID 34544504
- [Background] Zelen M. A new design for randomized clinical trials. N Engl J Med. 1979 May 31;300(22):1242-5. doi: 10.1056/NEJM197905313002203. PMID 431682
- [Background] Zelen M. Alternatives to classic randomized trials. Surg Clin North Am. 1981 Dec;61(6):1425-32. doi: 10.1016/s0039-6109(16)42596-x. PMID 7313934
- [Background] Zelen M. Randomized consent designs for clinical trials: an update. Stat Med. 1990 Jun;9(6):645-56. doi: 10.1002/sim.4780090611. PMID 2218168
- [Background] Torgerson DJ, Roland M. What is Zelen's design? BMJ. 1998 Feb 21;316(7131):606. doi: 10.1136/bmj.316.7131.606. No abstract available. PMID 9518917
- [Background] Peterson LR, Xanthakis V, Duncan MS, Gross S, Friedrich N, Volzke H, Felix SB, Jiang H, Sidhu R, Nauck M, Jiang X, Ory DS, Dorr M, Vasan RS, Schaffer JE. Ceramide Remodeling and Risk of Cardiovascular Events and Mortality. J Am Heart Assoc. 2018 May 3;7(10):e007931. doi: 10.1161/JAHA.117.007931. PMID 29728014